CLINICAL TRIAL: NCT00748995
Title: CSP #566 - Neuropsychological and Mental Outcomes of Operation Iraqi Freedom (OIF): A Longitudinal Cohort Study
Brief Title: Neuropsychological and Mental Outcomes of Operation Iraqi Freedom (OIF): A Longitudinal Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 566
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: None Retained — No Biospecimens were collected
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Neurocognition Deployment Health Study (NDHS) participants: Surviving NDHS participants who returned from their initial deployment to Iraq or Afghanistan.

SUMMARY:
This is a research study examining health effects of the Iraq War, especially those effects involving mental health. This study is a follow-up to the Neurocognition Deployment Health Study (NDHS), also called "Prospective Assessment of Neurocognition in Future Gulf-deployed and Gulf-nondeployed Military Personnel: A Pilot Study." The specific purpose of this research study is to find out more about the longer lasting effects of war on mood and stress symptoms, thinking and reaction skills, and different aspects of day to day life, such as work and daily activities. Survey and test results from previous participation in the NDHS will be compared to the new information that will be obtained from participants as part of this study. The investigators expect that a total of about 817 military personnel and military Veterans will participate in the study. There are two parts to this study: (1) mail/internet/phone survey and (2) in-person assessment. The investigators will invite all NDHS participants who deployed to Iraq to participate in the survey component. The survey component of the study involves being interviewed by phone about mood and stress symptoms and head injuries and completing written survey questions by either mail or on the internet that address basic personal history (such as age, military status, gender, combat injury history), mood, stress symptoms, and stressful experiences. The phone interview will take about 2 to 2.5 hours to complete. The questionnaire part will take about 20 to 30 minutes to complete, and can be completed either by mailing back completed questionnaires or by internet using a private, individual log-in/password combination. The investigators will invite approximately 200 selected at random from the larger group of survey responders to take part in the in-person assessment. The in-person assessment involves taking a small subset of neuropsychological tasks. The tasks will be given on a computer or using paper and pencil. Participants will also be asked to complete questionnaires about work, daily activities, and health history, as well as basic health measures such as height, weight, blood pressure, heart rate, and waist size. Potential participants will be given the option of completing the in-person assessment at one of the two study sites (Seattle or Boston), or in a private setting in their community (e.g., a hotel small conference room). Altogether, this part of the study will take about 120 minutes to 140 minutes to complete.

DETAILED DESCRIPTION:
As of August 2007, approximately 1.5 million U.S. service members had been deployed to either Iraq (Operation Iraqi Freedom, OIF) or Afghanistan (Operating Enduring Freedom, OEF). The sacrifices of these service members include >3500 fatalities and >35,000 injuries resulting in medical air transports. Medical sequelae, such as those involving traumatic amputations and traumatic brain injury, have been common. Contemporary military operations have also been linked to significant adverse mental health consequences. In particular, recent evidence suggests that both overt psychiatric symptoms and other functionally-relevant problems, such as attention and memory impairment, occur. These adverse mental health consequences, already observed in the immediate aftermath of war, could constitute a significant public health problem if prevalent and persistent.

In this context, Cooperative Studies Program (CSP) study #566 proposes an observational cohort design to examine war-related mental health dysfunction beyond the immediate aftermath of war. The proposed work builds on a unique data set available from the Neurocognition Deployment Health Study (NDHS), an interagency collaboration between the Department of Defense (DoD) and the Department of Veterans Affairs (VA). Initiated in April 2003, with an initial enrollment of 1595 participants, the NDHS has focused on short-term mental health outcomes of OIF deployment. To date, the NDHS is the only deployment health study of U.S. troops that includes both prospectively-gathered pre-deployment (baseline) and post-deployment (within 90 days after return from the war) data, as well as objective, performance-based measures of mental functioning.

The proposed work would collect new "long-term follow-up" data 3 to 5 years after NDHS participants returned from their initial deployment to Iraq. The newly acquired data from the proposed work will be analyzed with data available from the previous waves of the NDHS. The two primary objectives of CSP #566 are to: (1) determine the prevalence and course of posttraumatic stress disorder (PTSD) among Iraq War Veterans 3-5 years following return from their Iraq War deployment; and (2) assess the persistence of previously observed neuropsychological changes (in attention, verbal learning, visual memory, and reaction time) following war-zone participation and their relationships to the subsequent development of PTSD as the end-point. The second primary objective also evaluates traumatic brain injury (TBI) as a possible neural risk factor for PTSD.

The two secondary objectives are to: (1) examine the association of risk and resilience factors, including the impact of war zone stressors, with the outcomes of PTSD, major depressive disorder (MDD), and panic disorder; and (2) determine whether changes in PTSD symptoms or neuropsychological function are associated with subsequent day-to-day functioning, including health-related functional activities and occupational functioning.

The proposed study includes two hierarchical participant sampling frames: (1) a "full sample" (N=817) for examination of PTSD and related outcomes; and (2) a "neuropsychological subsample" (N=200) for examination of neuropsychological and functional outcomes. Both samples are drawn from the anticipated 1149 participants from the original NDHS cohort who deployed to Iraq and consented to be contacted for future research. The "full sample" component includes clinician-administered structured psychiatric phone interviews to determine clinically significant cases of PTSD, major depressive disorder, and panic disorder; a mail questionnaire survey will provide assessment of posttraumatic stress (PTS) symptom severity. The "neuropsychological sample" component includes in-person performance-based assessment of neuropsychological outcomes, shown previously to be affected by deployment to Iraq. In addition, participants in the neuropsychological sample will complete questionnaires relevant to health-related functional impact and occupational functioning.

The planned duration of the study is 5.5 years, including a 6 month start-up period, 42 months to locate, contact, and complete assessments on participants, 6 months to lock and close the database, and 12 months to complete the primary and secondary analyses. The attributes of the established study population, in combination with the scope of the proposed work, offer a unique opportunity to answer scientific questions with direct relevance to healthcare policy for returning OIF Veterans. Specifically, this study can 1) identify quantifiable and objective measures associated with subsequent outcome and functioning, 2) determine early potentially modifiable factors that may be used to promote resilience, 3) optimize treatment "windows," and 4) help project future resource allocation based on the frequency and impact of the mental health problems identified.

ELIGIBILITY:
Inclusion Criteria:

* Deployment to Iraq with completed NDHS baseline assessments

Exclusion Criteria:

* non-deployed,
* sensory-motor or cognitive loss sufficiently profound to permit meaningful participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surviving members of the NDHS cohort of 1595 participants
Sampling Method: Non-Probability Sample
Enrollment: 817 (Actual)
Dates: Start 2010-08-31 (Actual); Primary Completion 2014-07-10 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
PTSD diagnosis (current CAPS dx); PTSD threshold (PCL derived screening estimate) | 5 years
  1. PTSD dx (current CAPS dx at T3)
  2. PTSD threshold dx (PCL-derived screening estimate) for T3 vs. T1 comparison
  3. Trajectory patterns of PTSD threshold dx* (PCL-derived screening estimate) at T1, T2, and/or T3:
     * never (T1-,T2-,T3-)
     * persistent (T1-,T2+,T3+)
     * recovered (T1-,T2+,T3-)
     * late onset (T1-,T2-,T3+)
     * all others, e.g., pre- existing (T1+,T2+,T3+)
  [* +/- regarding PTSD threshold at time T1,2,3]
Neuropsych performance | 5 years
  * Neuropysch performance (T1 v. T2 v. T3)
  * PTSD diagnosis (CAPS dx); PTS symptom severity (PCL summary scores) (T3)

SECONDARY OUTCOMES:
Association of early/deploy/post-deploy stress exposures and PTSD, MDD, panic | 5 years
  * PTSD (CAPS current dx) (T3)
  * Mood Disorders, Panic Disorder, Agoraphobia, and Generalized Anxiety Disorders (MINI) (T3)
  * PTS symptom severity (PCL summary scores) (T3)
  * Depression symptom severity (CES-D summary scores) (T3)
  * Anxiety symptoms severity (DASS anxiety subscale) (T3)
Association from pre-deploy to long-term follow-up (T3) | 5 years
  * Employment (T3)
  * Absenteeism (HPQ) (T3)
  * Work performance (HPQ) (T3)
  * Health-related functioning (SFv12) (T3)
  * Cognitive-related functioning (MOS CF) (T3)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J Vasterling, PhD, Study Chair — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (4):
- United States (4):
  - CERC (VISN1, West Haven, CT), West Haven, Connecticut
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vasterling JJ, Aslan M, Proctor SP, Ko J, Marx BP, Jakupcak M, Schnurr PP, Gleason T, Huang GD, Concato J. Longitudinal Examination of Posttraumatic Stress Disorder as a Long-Term Outcome of Iraq War Deployment. Am J Epidemiol. 2016 Dec 1;184(11):796-805. doi: 10.1093/aje/kww151. Epub 2016 Nov 16. PMID 27852604
- [Result] Alosco ML, Aslan M, Du M, Ko J, Grande L, Proctor SP, Concato J, Vasterling JJ. Consistency of Recall for Deployment-Related Traumatic Brain Injury. J Head Trauma Rehabil. 2016 Sep-Oct;31(5):360-8. doi: 10.1097/HTR.0000000000000201. PMID 26580696
- [Result] Vasterling JJ, Aslan M, Lee LO, Proctor SP, Ko J, Jacob S, Concato J. Longitudinal Associations among Posttraumatic Stress Disorder Symptoms, Traumatic Brain Injury, and Neurocognitive Functioning in Army Soldiers Deployed to the Iraq War. J Int Neuropsychol Soc. 2018 Apr;24(4):311-323. doi: 10.1017/S1355617717001059. Epub 2017 Dec 4. PMID 29199924
- [Result] Aslan M, Concato J, Peduzzi PN, Proctor SP, Schnurr PP, Marx BP, McFall M, Gleason T, Huang GD, Vasterling JJ. Design of "neuropsychological and mental health outcomes of operation Iraqi freedom: a longitudinal cohort study". J Investig Med. 2013 Mar;61(3):569-77. doi: 10.2310/JIM.0b013e31828407ff. PMID 23392054
- [Result] Vasterling JJ, Proctor SP, Aslan M, Ko J, Jakupcak M, Harte CB, Marx BP, Concato J. Military, demographic, and psychosocial predictors of military retention in enlisted army soldiers 12 months after deployment to Iraq. Mil Med. 2015 May;180(5):524-32. doi: 10.7205/MILMED-D-14-00468. PMID 25939106
- [Result] Vasterling JJ, Aslan M, Proctor SP, Ko J, Leviyah X, Concato J. Long-term negative emotional outcomes of warzone TBI. Clin Neuropsychol. 2020 Aug;34(6):1088-1104. doi: 10.1080/13854046.2020.1749935. Epub 2020 Apr 17. PMID 32301397
- [Result] Jackson CE, Ciarleglio MM, Aslan M, Marx BP, Ko J, Concato J, Proctor SP, Vasterling JJ. Associations Among Increases in Posttraumatic Stress Symptoms, Neurocognitive Performance, and Long-Term Functional Outcomes in U.S. Iraq War Veterans. J Trauma Stress. 2021 Jun;34(3):628-640. doi: 10.1002/jts.22663. Epub 2021 Mar 2. PMID 33650202
- [Result] Vasterling JJ, Franz MR, Lee LO, Kaiser AP, Proctor SP, Marx BP, Schnurr PP, Ko J, Concato J, Aslan M. Early predictors of chronic posttraumatic stress disorder symptom trajectories in U.S. Army soldiers deployed to the Iraq war zone. J Trauma Stress. 2023 Oct;36(5):955-967. doi: 10.1002/jts.22964. Epub 2023 Aug 22. PMID 37608526
- See also: Related Info — http://www.research.va.gov/programs/csp/csp566.cfm
- See also: Related Info — http://www.research.va.gov/programs/csp/aslan-etal-2013.pdf